CLINICAL TRIAL: NCT07309939
Title: Effect of Gimkit-Based Gamified Learning on Achievement Motivation, Academic Performance, and Game Experience in Respiratory Skills Training: A Randomized Controlled Trial
Brief Title: Effect of Gimkit-Based Gamified Learning on Achievement Motivation, Academic Performance, and Game Experience in Respiratory Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Gamze Bolattürk, Assist. Prof., Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GİMKİT-RCT
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Gamified Learning; Gimkit; Game Based Learning; Nursing Students; Respiratory System Skills; Achievement Motivation; Academic Achievement; Gamification; Gamification in Health Education

STUDY DESIGN:
Who Masked: Participant
Masking Description: In the randomization process, those who meet the criteria for inclusion in the sample and accept to participate in the study do not know that they will be included in the intervention group or the control group, so it will be single-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gimkit Game-Based Learning (Experimental): The intervention planned for the study is a Gimkit-based game-enhanced learning method. Students in the experimental group participating in the respiratory system skills training will receive the standard skills laboratory instruction followed by a digital game session delivered through the Gimkit platform. The Gimkit activity includes interactive, competitive, and reinforcement-oriented questions designed to review key steps, principles, and safety considerations related to respiratory system procedures. The game session aims to increase student engagement, support recall, and enhance learning through gamification elements such as real-time feedback, point-based progression, and competition.
  Interventions: Behavioral: Gimkit Game-Based Learning
- Control Group (No Intervention): Students in the control group will receive only the standard respiratory system skills laboratory training, which includes instructor-led demonstration, supervised practice, and competency-based skills application. No game-based or digital reinforcement activity will be provided. After completing the laboratory session, students will take the same post-training multiple-choice knowledge test and post-intervention achievement motivation scale administered to the experimental group.

INTERVENTIONS:
Behavioral: Gimkit Game-Based Learning — The intervention consists of a game-enhanced learning session delivered through the Gimkit digital platform following the standard respiratory system skills laboratory training. The Gimkit activity includes interactive, competitive, and reinforcement-focused questions designed to review key knowledge and procedural steps related to respiratory system skills. Students receive immediate feedback, gain points, and experience gamified learning elements such as competition and real-time progress tracking. The session aims to increase engagement, enhance motivation, and support learning retention after the laboratory training. Duration of the intervention is approximately 20-30 minutes and is applied only once during the study period.
  Arms: Gimkit Game-Based Learning

SUMMARY:
This randomized controlled trial aims to examine the effect of Gimkit-based game-enhanced learning on achievement motivation, academic performance, and game experience among first-year nursing students during respiratory system skills training. Students are randomly assigned to either the experimental group, which receives standard respiratory skills laboratory training followed by a Gimkit game session designed to reinforce key concepts, or the control group, which receives only the standard skills laboratory training. Achievement motivation is assessed using the Expectancy-Value Theory-based Achievement Motivation Scale before and after the intervention in both groups. Academic performance is evaluated using a 10-item multiple-choice digital test administered after the skills laboratory session. Additionally, the Game Experience Scale is administered to students in the experimental group to measure their perceptions of game-based learning. The study aims to determine whether game-based reinforcement improves motivation and learning outcomes compared with traditional laboratory instruction.

DETAILED DESCRIPTION:
Nursing education increasingly incorporates digital and game-based strategies to enhance student engagement, motivation, and performance. Gimkit is an interactive, competitive, game-based learning platform shown to improve recall, engagement, and active learning.

In this study, nursing students enrolled in the Fundamentals of Nursing course receive training on respiratory system skills. The experimental group participates in a game-based reinforcement session using Gimkit immediately after the skills laboratory, whereas the control group receives only traditional skills laboratory training.

Measurements:

Achievement Motivation Scale (Expectancy-Value Theory-based, 9 items, 2 subscales): administered pre- and post-intervention for both groups.

Academic success test (10-item multiple-choice digital test): administered post-intervention to both groups.

Game Experience Scale (5 subdimensions): administered post-intervention to the experimental group only.

The study evaluates the effect of the Gimkit intervention on changes in motivation and academic achievement and explores students' game experience perceptions.

ELIGIBILITY:
Inclusion Criteria:

* First-year nursing students
* Enrolled in Fundamentals of Nursing course
* Participating in respiratory system skills laboratory
* Volunteering to participate in the study

Exclusion Criteria:

* Not attending the skills laboratory session
* Not completing pre- or post-tests

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Achievement Motivation Score | Pre-intervention (baseline) and immediately post-intervention
  Achievement motivation will be measured using the Expectancy-Value Theory-based Achievement Motivation Scale, which consists of 9 items and 2 subdimensions (Expectancy and Task Value). Each item is rated on a Likert scale, and higher scores indicate higher achievement motivation. The scale will be administered to both the experimental and control groups before and after the intervention. Results will be aggregated and reported as total score and subscale scores (mean ± standard deviation).
Academic Achievement (Knowledge Test Score) | Two weeks after the skills lab session
  Academic achievement will be measured using a 10-item multiple-choice digital test assessing knowledge related to respiratory system skills. Each correct answer is scored as 1 point, resulting in a total possible score of 0-10. Higher scores indicate better academic performance. The test will be administered to both groups immediately after the respiratory skills laboratory session. Results will be reported as mean ± standard deviation.

SECONDARY OUTCOMES:
Game Experience Score | Immediately post-intervention (after the Gimkit session)
  Students in the experimental group will complete the Game Experience Scale following the Gimkit session. The scale includes multiple subdimensions (e.g., engagement, enjoyment, flow, usability, perceived learning value). Items are rated on a Likert scale, and higher scores indicate a more positive game-based learning experience. Results will be aggregated for total and subdimension scores and reported as mean ± standard deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Üniversitesi, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No